CLINICAL TRIAL: NCT07357272
Title: A Cohort Study on Increasing Blood Pressure Benefits in Sleep Apnea Patients After CPAP Treatment
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025179
Record Dates: First submitted 2025-09-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Hypertension (HTN); Sleep Apnea Syndrome, Obstructive
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, feces, saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hypertension with OSA: We will enroll 200 adults 18-70 y with newly-diagnosed obstructive sleep apnea (AHI ≥5 + symptoms or ≥15/h) and untreated or sub-optimally controlled blood pressure (120-159/80-99 mmHg or on stable meds but not at target). All will undergo auto-titrating CPAP for 3 months (≥4 h/night, ≥21 nights/month) with mask-fitting, education and side-effect management to maximize adherence. Participants who report insomnia or frequent CPAP-related awakenings may additionally receive 4-week bedtime trazodone (25-150 mg) or zopiclone (3.75-7.5 mg) at physician discretion, creating natural sub-groups: CPAP-only, CPAP+trazodone, CPAP+zopiclone, or drug-only for those refusing CPAP. Outcomes: 24-h BP change, CPAP adherence, subjective/objective sleep quality. Exclusions: prior OSA therapy, secondary hypertension, unstable cardiopulmonary disease, pregnancy, rotating night shift, recent hypnotic use, or concurrent interventional trials.
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — All will undergo auto-titrating CPAP for 3 months (≥4 h/night, ≥21 nights/month) with mask-fitting, education and side-effect management to maximize adherence.

SUMMARY:
Research Title "Quadruple-Blind Randomized Controlled Trial of the Effect of CPAP on Blood Pressure in Patients with Sleep Apnea" Why are we conducting this study?

* Sleep apnea (OSA) is very common, affecting approximately one in every eight adults. It makes it more difficult to control blood pressure.
* Continuous Positive Airway Pressure (CPAP) is the preferred treatment, but the effect on blood pressure varies from person to person.
* We want to know: Which patients experience the greatest reduction in blood pressure with CPAP? Can adding a little sleep aid medication for those who have trouble sleeping or frequently wake up at night improve the effectiveness of CPAP and lead to better blood pressure control? Who will participate?
* 18-70 years old, diagnosed with obstructive sleep apnea, with snoring, gasping, or daytime sleepiness.
* High blood pressure or newly diagnosed with mild hypertension, or taking 1-2 blood pressure-lowering medications but not reaching the target.
* Able to wear the CPAP mask every night and willing to undergo 3-month follow-up.
* Pregnant women, those already using CPAP, those with a history of heart disease/stroke in the last 3 months, those working night shifts ≥ 3 nights/week, or those participating in other intervention trials are not eligible.

What will the study do? First, conduct a full-night sleep monitoring and 24-hour blood pressure monitoring to adjust the most suitable CPAP pressure for you.

Wear the CPAP mask for ≥ 4 hours every night, for a total of ≥ 21 days per month, for approximately 3 months.

If you often wake up at night or have insomnia, you can voluntarily join the "sleep aid medication" group: take trazodone (25-150 mg) or zolpidem (3.75-7.5 mg) before bedtime for 4 weeks.

During this period, we will use questionnaires, a small wristwatch (actigraphy), and additional sleep monitoring to observe changes in sleep and blood pressure; we will also draw a small amount of blood and collect urine for routine safety checks.

You can withdraw at any time without any penalty and it will not affect your regular medical treatment.

Possible benefits

* Free comprehensive assessment of sleep and blood pressure, one-on-one guidance from a doctor.
* May lead to a reduction in blood pressure and improvement in nighttime sleep quality.
* Help future patients like you receive better treatment. Possible discomfort or risks
* CPAP: mask pressure marks, dry mouth and nose, feeling of suffocation, bloating; most people's symptoms are relieved after adjusting the humidifier or mask.
* Sleep aid medication: next-day drowsiness, dry mouth, dizziness, nausea; rare cases may include persistent penile erection in men (immediate medical consultation required); the risk of dependency for zolpidem after continuous use for 4 weeks is very low, but it still requires monitoring by a doctor.
* Check: wearing a blood pressure cuff and sleep monitoring device may cause slight inconvenience during sleep.
* If there is any injury related to the study, Anzhen Hospital will provide necessary treatment and compensation in accordance with Chinese laws.

Privacy and Costs

* Sleep monitoring, dynamic blood pressure, medications, and tests required for the study are all free.
* Your name and medical record will only be viewed by researchers and the ethics committee. Personal identity will not be disclosed when the article is published. Contact person
* Research Question: Dr. Xie Jiang 010-64456528 (during working days) / 131-6198-5564 (at other times)
* Rights and Benefits: Beijing Anzhen Hospital Ethics Committee 010-64456214 Voluntary Decision Whether to participate or not is completely voluntary. You can withdraw at any time without any reason, and it will not affect the medical care you are entitled to.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years old;
2. Diagnosed with obstructive sleep apnea (OSA) through overnight polysomnography (PSG), as follows: (1) AHI ≥ 5 times/hour and one of the following conditions is met: (1) The patient complains of daytime sleepiness, lack of sleepiness during sleep, fatigue or insomnia; (2) Waking up due to breathlessness or wheezing; (3) The bed partner or other witnesses report that the patient has habitual snoring, breathing interruptions or both during sleep. Or (2) AHI ≥ 15 times/hour.
3. Satisfy any of the following blood pressure conditions: (1) Office blood pressure 120-139/80-89 mmHg, with ≤ 2 cardiovascular risk factors; (2) Newly diagnosed blood pressure 140-159/90-99 mmHg and without cardiovascular risk factors; (3) Currently taking stable types and doses of antihypertensive drugs, but the office blood pressure has not reached the normal blood pressure standard (120/80 mmHg) with a low-risk level of cardiovascular risk for patients with hypertension; (4) Any non-cardiovascular risk level high-risk patient who voluntarily requests three-month CPAP treatment and accepts follow-up;
4. Able to tolerate 24-hour ambulatory blood pressure monitoring and continuous blood pressure monitoring;

Exclusion Criteria:

1. Previously diagnosed with OSA and currently undergoing OSA treatment (such as CPAP, orthodontic devices, surgery, etc.);
2. Secondary hypertension caused by other reasons other than OSA, such as renal artery stenosis, kidney disease, Cushing's syndrome, primary aldosteronism;
3. Unstable condition (having experienced cardiovascular events or major surgeries in the past 3 months, severe sleepiness (ESS ≥ 16 points), or cognitive impairment that makes it impossible to cooperate, active mental illness or drug/alcohol abuse);
4. Rheumatic immune diseases and malignant tumors;
5. Large artery diseases (such as giant cell arteritis, arterial dissection, aneurysm, etc.);
6. Diseases that cannot accurately measure blood pressure (such as atrial fibrillation, upper limb vascular diseases);
7. Early-onset familial hypertension;
8. Any prescription or over-the-counter sleep aid (benzodiazepines, non-benzodiazepines, melatonin receptor agonists, trazodone, sedative antipsychotic/antidepressants containing sedative components, OTC containing sedative components) within 4 weeks before enrollment;
9. Allergic or contraindicated to the potential study drugs (trazodone, zopiclone);
10. Pregnant, lactating, or planning to become pregnant;
11. Frequent night shift work (≥ 3 nights/week) or circadian rhythm disorder (diagnosed by a doctor);
12. Participating in other interventional clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who meet the age and screening criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure | After 3 months of CPAP treatment
  The changes in blood pressure of the patient after receiving CPAP treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Currently, this trial is focused on completing the recruitment of participants and conducting the analysis of the primary endpoints. The final form and platform for data sharing have not yet been determined. Given that IPD sharing needs to take into account patient privacy protection, renewal of ethical approval, and negotiations regarding the intellectual property rights of the funding party, we reserve the right to formulate and upload a specific sharing plan (including de-identified data sets, analysis codes, and research protocols) within 6 months before the publication of the paper. Therefore, at this stage, we choose "Undecided". If we decide to share in the future, it will be freely accessible through OSF or a domestic compliant data repository in accordance with ICMJE requirements, and the registration record will be updated. If we ultimately do not share, the reasons will be clearly stated in this column.

REFERENCES:
- [Result] Meng Z, Chen Y, Yang T, Sun B, Luo C, Wei G, Xie X, Gu Y, Ding N, Zhang X, Xu J. New perspective on exploring the predictive factors of blood pressure reduction during CPAP treatment in people with severe OSA and hypertension: a prospective observational study. BMJ Open Respir Res. 2023 May;10(1):e001560. doi: 10.1136/bmjresp-2022-001560. PMID 37169401
- [Result] Pengo MF, Oscullo G, Gomez-Olivas JD, Bilo G, Parati G, Martinez-Garcia MA. Nocturnal BP Profile Predicts CPAP Effect on BP in Patients With OSA and Resistant Hypertension. Chest. 2023 Nov;164(5):1302-1304. doi: 10.1016/j.chest.2023.05.021. Epub 2023 Jun 17. No abstract available. PMID 37364854
- [Result] Sanchez-de-la-Torre M, Gracia-Lavedan E, Benitez ID, Zapater A, Torres G, Sanchez-de-la-Torre A, Aldoma A, de Batlle J, Targa A, Abad J, Duran-Cantolla J, Urrutia A, Mediano O, Masdeu MJ, Ordax-Carbajo E, Masa JF, De la Pena M, Mayos M, Coloma R, Montserrat JM, Chiner E, Minguez O, Pascual L, Cortijo A, Martinez D, Dalmases M, Lee CH, McEvoy RD, Barbe F; Spanish Sleep Network. Long-Term Effect of Obstructive Sleep Apnea and Continuous Positive Airway Pressure Treatment on Blood Pressure in Patients with Acute Coronary Syndrome: A Clinical Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1750-1759. doi: 10.1513/AnnalsATS.202203-260OC. PMID 35442180
- [Result] Labarca G, Schmidt A, Dreyse J, Jorquera J, Enos D, Torres G, Barbe F. Efficacy of continuous positive airway pressure (CPAP) in patients with obstructive sleep apnea (OSA) and resistant hypertension (RH): Systematic review and meta-analysis. Sleep Med Rev. 2021 Aug;58:101446. doi: 10.1016/j.smrv.2021.101446. Epub 2021 Jan 28. PMID 33607443
- [Result] Wu H, Guo Y. Risk of resistant hypertension associated with insomnia in patients with obstructive sleep apnea. Sleep Med. 2023 Jan;101:445-451. doi: 10.1016/j.sleep.2022.12.001. Epub 2022 Dec 5. PMID 36516601
- [Result] Shiina K. Obstructive sleep apnea -related hypertension: a review of the literature and clinical management strategy. Hypertens Res. 2024 Nov;47(11):3085-3098. doi: 10.1038/s41440-024-01852-y. Epub 2024 Aug 29. PMID 39210083

DOCUMENTS (2):
  • Study Protocol (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT07357272/Prot_000.pdf
  • Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT07357272/ICF_001.pdf